CLINICAL TRIAL: NCT06340581
Title: A Phase I, Randomized, Partial Double-blind, Single Dose, 3 Way Cross Over Study to Assess the Lung Exposure Bioequivalence of Budesonide, Glycopyrronium, and Formoterol for BGF MDI HFO Compared With BGF MDI HFA Using an AeroChamber Plus Flow Vu Spacer and to Compare the Lung Exposure of BGF MDI HFO With a Spacer to BGF MDI HFO Without a Spacer
Brief Title: A Study to Assess the Lung Exposure Bioequivalence of Budesonide, Glycopyrronium, & Formoterol (BGF) Metered Dose Inhaler (MDI) With a Next-generation Propellant (NGP) With a Spacer, BGF MDI Hydrofluoroalkane (HFA) With a Spacer, as Well as BGF MDI NGP Without a Spacer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study no longer required.
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5985C00009; 2023-509914-12 (Other: EU CT)
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Ex-actuator; AeroChamber; Spacer; COPD with moderate to severe airflow obstruction; Long-acting beta2-agonist (LABA); Long-acting muscarinic antagonist (LAMA); Propellant; Next Generation Propellant (NGP); Inhaled Corticosteroid (ICS); Lung Exposure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (6):
- Treatment Sequence 1: ABC (Experimental): Participants will be randomized to one of the 6 different treatment sequences. Each participant will receive single-dose treatments of BGF MDI HFA with spacer (Treatment A), followed by BGF MDI HFO with spacer (Treatment B), and then BGF MDI HFO without spacer (Treatment C) in 3 treatment periods with single dose (4 puffs) on Day 1 of all treatment periods.
  Interventions: Drug: Treatment A: BGF MDI HFA; Drug: Treatment B: BGF MDI HFO; Drug: Treatment C: BGF MDI HFO; Device: AeroChamber Plus Flow-Vu Spacer
- Treatment Sequence 2: ACB (Experimental): Participants will be randomized to one of the 6 different treatment sequences. Each participant will receive single-dose treatments of BGF MDI HFA with spacer (Treatment A), followed by BGF MDI HFO without spacer (Treatment C), and then BGF MDI HFO with spacer (Treatment B) in 3 treatment periods with single dose (4 puffs) on Day 1 of all treatment periods.
  Interventions: Drug: Treatment A: BGF MDI HFA; Drug: Treatment B: BGF MDI HFO; Drug: Treatment C: BGF MDI HFO; Device: AeroChamber Plus Flow-Vu Spacer
- Treatment Sequence 3: BAC (Experimental): Participants will be randomized to one of the 6 different treatment sequences. Each participant will receive single-dose treatments of BGF MDI HFO with spacer (Treatment B), followed by BGF MDI HFA with spacer (Treatment A), and then BGF MDI HFO without spacer (Treatment C) in 3 treatment periods with single dose (4 puffs) on Day 1 of all treatment periods.
  Interventions: Drug: Treatment A: BGF MDI HFA; Drug: Treatment B: BGF MDI HFO; Drug: Treatment C: BGF MDI HFO; Device: AeroChamber Plus Flow-Vu Spacer
- Treatment Sequence 4: BCA (Experimental): Participants will be randomized to one of the 6 different treatment sequences. Each participant will receive single-dose treatments of BGF MDI HFO with spacer (Treatment B) followed by BGF MDI HFO without spacer (Treatment C), and then BGF MDI HFA with spacer (Treatment A) in 3 treatment periods with single dose (4 puffs) on Day 1 of all treatment periods.
  Interventions: Drug: Treatment A: BGF MDI HFA; Drug: Treatment B: BGF MDI HFO; Drug: Treatment C: BGF MDI HFO; Device: AeroChamber Plus Flow-Vu Spacer
- Treatment Sequence 5: CAB (Experimental): Participants will be randomized to one of the 6 different treatment sequences. Each participant will receive single-dose treatments of BGF MDI HFO without spacer (Treatment C), followed by BGF MDI HFA with spacer (Treatment A), and then BGF MDI HFO with spacer (Treatment B) in 3 treatment periods with single dose (4 puffs) on Day 1 of all treatment periods.
  Interventions: Drug: Treatment A: BGF MDI HFA; Drug: Treatment B: BGF MDI HFO; Drug: Treatment C: BGF MDI HFO; Device: AeroChamber Plus Flow-Vu Spacer
- Treatment Sequence 6: CBA (Experimental): Participants will be randomized to one of the 6 different treatment sequences. Each participant will receive single-dose treatments of BGF MDI HFO without spacer (Treatment C), followed by BGF MDI HFO with spacer (Treatment B), and then BGF MDI HFA with spacer (Treatment A) in 3 treatment periods with single dose (4 puffs) on Day 1 of all treatment periods.
  Interventions: Drug: Treatment A: BGF MDI HFA; Drug: Treatment B: BGF MDI HFO; Drug: Treatment C: BGF MDI HFO; Device: AeroChamber Plus Flow-Vu Spacer

INTERVENTIONS:
Drug: Treatment A: BGF MDI HFA — Participants will receive 4 oral inhalations of BGF MDI HFA as a single dose with AeroChamber Plus Flow-Vu spacer with charcoal.
Drug: Treatment B: BGF MDI HFO — Participants will receive 4 oral inhalations of BGF MDI HFO as a single dose with AeroChamber Plus Flow-Vu spacer with charcoal.
Drug: Treatment C: BGF MDI HFO — Participants will receive 4 oral inhalations of BGF MDI HFO as a single dose without spacer with charcoal.
Device: AeroChamber Plus Flow-Vu Spacer — Participants will receive 4 inhalations of BGF MDI HFA (treatment A) and BGF MDI HFO (Treatment B) as a single dose with AeroChamber Plus Flow-Vu spacer.

SUMMARY:
The primary purpose of this study is to demonstrate the equivalence of budesonide, glycopyrronium, formoterol (BGF) metered dose inhaler (MDI) hydrofluoroolefin (HFO) with a spacer to BGF MDI hydrofluoroalkane (HFA) with a spacer. The secondary objective is to characterize BGF MDI HFO with and without a spacer.

DETAILED DESCRIPTION:
This study is a Phase I, randomized, partial double-blind, single dose, single-center, 3-way cross over study to assess the pharmacokinetic (PK) and safety of BGF MDI in healthy participants (male or female).

The study will comprise:

1. A Screening Period of up to 27 days prior to first dosing.
2. Three treatment periods: Participants will be resident at the Clinical Unit from Day -1 until 24 hours after dosing with the final treatment.
3. Follow-up: A final Follow-up Phone Call within 5 to 7 days after the last administration of BGF MDI in Treatment Period 3.

Participants will receive all 3 treatments as a single dose (4 inhalations) (Treatment A [BGF MDI HFA with AeroChamber Plus Flow-Vu spacer with charcoal, reference formulation], Treatment B [BGF MDI HFO with AeroChamber Plus Flow-Vu spacer with charcoal - test formulation], and Treatment C [BGF MDI HFO without spacer with charcoal]) (1 treatment per treatment period) in one of 6 possible treatment sequences; ABC, ACB, BAC, BCA, CAB, or CBA.

There will be a 3 to 7 days washout period between each dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Females must have a negative pregnancy test at screening and on admission to the Clinical Unit, must not be lactating.
* Have a body mass index (BMI) between 18 and 30 kilograms per meter square (kg/m^2) inclusive and weigh at least 50 kilograms (kg).
* Have a FEV1 greater than or equal to (>=) 80 percentage (%).
* Demonstrate basic understanding of how to use an MDI device with and without a spacer after receiving training.
* Participants should be fully/sufficiently vaccinated as per local definitions against severe acute respiratory syndrome coronavirus type 2 (SARS CoV-2).

Exclusion Criteria:

* History or current evidence of any clinically significant disease or disorder, including endocrinological diseases, such as thyrotoxicosis, which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the results through participation in the study.
* History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational medicinal product (IMP).
* History of narrow angle glaucoma or change in vision.
* History of symptomatic prostatic hypertrophy or bladder neck obstruction/urinary retention.
* Unresectable cancer that has not been in complete remission for at least 5 years.
* Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results.
* Any clinically significant abnormal findings in physical examination or vital signs at screening, as judged by the investigator. Eg., Systolic blood pressure (BP) less than (<) 90 millimeters of Mercury (mmHg) or greater than or equal to (>=) 140 mmHg and diastolic BP < 50 mmHg or >=90 mmHg; Heart rate < 50 beats per minute (bpm) or > 90 bpm.
* Any clinically significant abnormalities on 12-lead electrocardiogram (ECG) at screening, as judged by the investigator.
* Any positive result on screening for serum hepatitis B surface antigen (HBsAg) OR anti-hepatitis B core (HBc) antibody, indicative of hepatitis B, hepatitis C antibody, or human immunodeficiency virus (HIV).
* Positive reverse transcription polymerase chain reaction (RT-PCR) test for SARS-CoV-2 prior to randomization.
* Participant has clinical signs and symptoms consistent with Coronavirus disease 2019 (COVID-19), eg, fever, dry cough, dyspnea, sore throat, fatigue, new smell or taste disorder or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or on admission.
* Participant who had severe course of COVID-19 (ie, hospitalization, extracorporeal membrane oxygenation, or mechanically ventilated).
* Recent (within 14 days prior to admission to the Clinical Unit) exposure to someone who has COVID-19 symptoms or tested positive for SARS-CoV-2.
* History of any respiratory disorders such as asthma, Chronic obstructive pulmonary disease (COPD), or idiopathic pulmonary fibrosis.
* Known or suspected history of drug abuse, as judged by the investigator.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days or 5 half-lives (whichever is longest) of the first administration of IMP in this study.
* Plasma donation within one month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity to drugs with a similar chemical structure or class to BGF or to its excipients, such as norflurane.
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months prior to screening.
* Positive screen for drugs of abuse or cotinine at screening or on admission to the Clinical Unit or positive screen for alcohol at screening or on admission to the Clinical Unit.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
* Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the investigator. Excessive intake of alcohol defined as the regular consumption of more than 24 g of alcohol per day for men or 12 g of alcohol per day for women.
* Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, chocolate).
* Participants who have previously received BGF MDI HFO.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-17 (Estimated); Primary Completion 2025-02-27 (Estimated); Study Completion 2025-02-27 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-curve from Zero to the Last Quantifiable Concentration (AUClast) of BGF MDI | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  The bioequivalence of the lung exposure of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO with a spacer compared with BGF MDI HFA with a spacer will be assessed.
Maximum Observed Concentration (Cmax) of BGF MDI | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  The bioequivalence of the lung exposure of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO with a spacer compared with BGF MDI HFA with a spacer will be assessed.

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-curve from Zero to the Last Quantifiable Concentration (AUClast) | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  The relative lung bioavailability of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO with a spacer versus BGF MDI HFO without a spacer will be assessed.
Maximum Observed Concentration (Cmax) | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  The relative lung bioavailability of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO with a spacer versus BGF MDI HFO without a spacer will be assessed.
Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf) | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  The lung exposure PK parameters of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO (with and without spacer) and BGF MDI HFA with a spacer will be assessed.
Time to Reach Maximum Observed Concentration (tmax) | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  The lung exposure PK parameters of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO (with and without spacer) and BGF MDI HFA with a spacer will be assessed.
Terminal Rate Constant (λz) | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  The lung exposure PK parameters of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO (with and without spacer) and BGF MDI HFA with a spacer will be assessed.
Half-life Associated with Terminal Slope (λz) of a Semi-logarithmic Concentration-time Curve (t1/2λz) | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  The lung exposure PK parameters of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO (with and without spacer) and BGF MDI HFA with a spacer will be assessed.
Mean Residence Time of the Unchanged Drug in the Systemic Circulation from Zero to Infinity (MRTinf) | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  The lung exposure PK parameters of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO (with and without spacer) and BGF MDI HFA with a spacer will be assessed.
Apparent Total Body Clearance of Drug from Plasma After Extravascular Administration (CL/F) | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  The lung exposure PK parameters of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO (with and without spacer) and BGF MDI HFA with a spacer will be assessed.
Apparent Volume of Distribution at Steady State Following Extravascular Administration (Vz/F) | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  The lung exposure PK parameters of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO (with and without spacer) and BGF MDI HFA with a spacer will be assessed.
Number of Participants with Adverse Events | From Baseline up to 48 days
  The safety and tolerability of single doses of BGF MDI HFO (with and without spacer) and BGF MDI HFA with a spacer, in healthy participants will be evaluated.

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment athttps://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/